CLINICAL TRIAL: NCT04473092
Title: Prospective Analysis of the Feasibility of the PASCAL Spacer Technology for Transcatheter Mitral Valve Repair in an All-comers Cohort
Acronym: OneForAll
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Peter Lüdike, Prof. Dr., University Hospital, Essen
Other Study IDs: 20-9223-BO
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: TMVR — Patients who undergo TMVR for MR at the PI´s site

SUMMARY:
To identify changes on mitral valve morphology and functionality by the application of the PascalTM in MR.

DETAILED DESCRIPTION:
Transcatheter mitral valve repair (TMVR) in mitral regurgitation (MR) is increasingly applied in patients on high surgical risk. Interventional mitral valve repair can be applied is routinely applied in primary and secondary mitral regurgitation. While the edge-to-edge technique has been the solely available technlology in the marked for the last years, the recently introduced PascalTM technology represents a novel concept and is characterized by a central spacer, wider paddles, and larger dimensions. Implications of implantation of the PascalTM device on the mitral valve morphology and functionality concerning potential changes on mitral regurgitation as well as changes on mitral valve orifice area are to date not fully understood. The current study will identify anatomical changes to optimize ideal patient selection and optimal treatment approaches of the PASCALTM device.

ELIGIBILITY:
Inclusion Criteria:

• All patients who undergo TVMR for MR (age >18yrs) at the PI´s site

Exclusion Criteria:

* <18yry
* Subject does not provide full consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo TVMR for MR (age >18yrs) at the PI´s site
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Morphologic and functional changes of mitral valve anatomy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lüdike, MD, Principal Investigator — University Hospital Essen, Westgerman Heart- and Vascular Center, Department of Cardiology and Vascular Medicine
Locations (1):
- University Hospital Essen, Westgerman Heart and Vascular Center, Department of Cardiology and Vascular Medicine, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No